CLINICAL TRIAL: NCT00000585
Title: Penicillin Prophylaxis in Sickle Cell Disease (PROPS)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Prevention
Other Study IDs: 305
Record Dates: First submitted 1999-10-27; First posted 1999-10-28 (Estimated); Last update posted 2016-03-25 (Estimated); Status verified 1994-10

CONDITIONS: Anemia, Sickle Cell; Hematologic Diseases; Hemoglobinopathies; Infection (S. Pneumoniae); Pneumonia
MeSH Terms: conditions — Anemia, Sickle Cell; Hematologic Diseases; Hemoglobinopathies; Infections; Pneumonia | interventions — Penicillins

INTERVENTIONS:
Drug: penicillin

SUMMARY:
To determine whether the regular daily administration of oral penicillin would reduce the incidence of documented infection due to Streptococcus pneumoniae in children with sickle cell anemia.

DETAILED DESCRIPTION:
BACKGROUND:

For over 20 years children with sickle cell anemia have been known to have an increased susceptibility to severe bacterial infection, particularly due to Streptococcus pneumoniae. Meningitis, pneumonia and septicemia due to this organism have been recognized as the major causes of death for these children, with children under three years of age being at highest risk. The annual incidence of pneumococcal septicemia among young children with sickle cell anemia appears to have remained remarkably constant over the last two decades at approximately 10 percent. This illness can often be fulminant, progressing from the onset of fever to death in less than 12 hours, with a case fatality rate ranging as high as 35 percent.

Penicillin prophylaxis has been advocated as a preventive measure against severe pneumococcal infections in children with sickle cell anemia. One study had shown that the risk of pneumococcal infection in these children could be reduced by the use of parenteral penicillin.

DESIGN NARRATIVE:

Phase I was a multi-center, randomized, double-blind, placebo-controlled trial. One hundred and five patients were assigned to the penicillin group and 110 to placebo. The primary endpoint was a documented severe infection due to S. pneumoniae. The secondary endpoint was a severe infection due to an organism other than S. pneumoniae.

Because data were not available to define the age at which prophylactic penicillin could be safely discontinued, the NHLBI launched Phase II of the Prophylactic Penicillin Study beginning in 1987. Recruitment ended in August, 1993. The clinical phase of Phase II ended in August, 1994.

Phase II was a multi-center randomized trial to evaluate the hazards of discontinuing daily oral penicillin at the age of five years. Within three months of their fifth birthdays, all children were randomized to continue oral penicillin prophylaxis or to stop prophylaxis. Each child was followed for a minimum of two years. The primary endpoint was a comparison of documented pneumococcal infection in children continuing penicillin after five years of age versus children whose prophylaxis was stopped at five years of age. Ancillary studies conducted in subsets of patients included: the prevalence of colonization of the nasopharynx with antibiotic resistant microorangisms; and the relationship of antibody response to pneumococcal vaccination to the incidence of pneumococcal sepsis in this patient population.

ELIGIBILITY:
In the Phase I trial, Black children with sickle cell anemia aged 3 months to 3 years. In the Phase II trial, children with sickle cell anemia aged five years 3 months of age and younger who had received prophylactic penicillin for at least two yea

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Dates: Start 1983-08; Study Completion 1994-10

CONTACTS AND LOCATIONS:
Overall Officials: David Becton — University of Arkansas; Ann Bjornson — Gamble Institute of Medical Research; George Buchanan — University of Texas; Neil Grossman — Children's Hospital Medical Center, Cincinnati; C. Holbrook — East Carolina University School of Medicine; Rathyi Iyer — University of Mississippi Medical Center; Karen Kalinyak — Children's Hospital Medical Center, Cincinnati; Thomas Kinney — Duke University; Helen Maurer — University of Illinois at Chicago; Scott Miller — New York Health Science Center; Charles Pegelow — University of Miami; Sergio Piomelli — Columbia University; Gregory Reaman — Children's Hospital National Medical Center; Alan Schwartz — Washington University School of Medicine; Elliott Vichinsky — Children's Hospital & Medical Center; Winfred Wang — St. Jude Children's Research Hospital; Doris Wethers — St. Luke's Roosevelt Institute of Health Science; Gerald Woods — Children's Mercy Hospital Kansas City

REFERENCES:
- [Background] Gaston MH, Verter JI, Woods G, Pegelow C, Kelleher J, Presbury G, Zarkowsky H, Vichinsky E, Iyer R, Lobel JS, et al. Prophylaxis with oral penicillin in children with sickle cell anemia. A randomized trial. N Engl J Med. 1986 Jun 19;314(25):1593-9. doi: 10.1056/NEJM198606193142501. PMID 3086721
- [Background] Falletta JM, Woods GM, Verter JI, Buchanan GR, Pegelow CH, Iyer RV, Miller ST, Holbrook CT, Kinney TR, Vichinsky E, et al. Discontinuing penicillin prophylaxis in children with sickle cell anemia. Prophylactic Penicillin Study II. J Pediatr. 1995 Nov;127(5):685-90. doi: 10.1016/s0022-3476(95)70154-0. PMID 7472817
- [Background] Bjornson AB, Falletta JM, Verter JI, Buchanan GR, Miller ST, Pegelow CH, Iyer RV, Johnstone HS, DeBaun MR, Wethers DL, Wang WC, Woods GM, Holbrook CT, Becton DL, Kinney TR, Reaman GH, Kalinyak K, Grossman NJ, Vichinsky E, Reid CD. Serotype-specific immunoglobulin G antibody responses to pneumococcal polysaccharide vaccine in children with sickle cell anemia: effects of continued penicillin prophylaxis. J Pediatr. 1996 Dec;129(6):828-35. doi: 10.1016/s0022-3476(96)70026-4. PMID 8969724
- [Background] Woods GM, Jorgensen JH, Waclawiw MA, Reid C, Wang W, Pegelow CH, Rogers ZR, Iyer RV, Holbrook CT, Kinney TR, Vichinsky E, DeBaun MR, Grossman NJ, Thomas MD, Falletta JM. Influence of penicillin prophylaxis on antimicrobial resistance in nasopharyngeal S. pneumoniae among children with sickle cell anemia. The Ancillary Nasopharyngeal Culture Study of Prophylactic Penicillin Study II. J Pediatr Hematol Oncol. 1997 Jul-Aug;19(4):327-33. doi: 10.1097/00043426-199707000-00011. PMID 9256832
- [Background] Gaston MH, Verter J. Sickle cell anaemia trial. Stat Med. 1990 Jan-Feb;9(1-2):45-9; discussion 49-51. doi: 10.1002/sim.4780090111. PMID 2111933